CLINICAL TRIAL: NCT01322269
Title: A Randomized, Open-Label, Multi-Dose Study of HQK-1001 in Subjects With Sickle Cell Disease
Brief Title: A Study of HQK-1001 in Patients With Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HemaQuest Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HQP 1001-SCD-006
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia; Sickle Cell Disorders; Hemoglobin S Disease; Sickling Disorder Due to Hemoglobin S
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — 2,2-dimethylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HQK-1001 (30 mg/kg) (Experimental)
  Interventions: Drug: HQK-1001
- HQK-1001 (40 mg/kg) (Experimental)
  Interventions: Drug: HQK-1001
- HQK-1001 (50 mg/kg) (Experimental)
  Interventions: Drug: HQK-1001

INTERVENTIONS:
Drug: HQK-1001 — HQK-1001 tablets, once daily for daily 26 weeks

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of three dose levels of HQK-1001 administered once daily for 26 weeks in subjects with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of SCD
* Males and females between 12 and 60 years of age, inclusive
* At least 3 episodes of a SCD-related crisis or complication in the 3 years prior to screening OR 1 episode of acute chest syndrome in the 5 years prior to screening
* If receiving hydroxyurea, must be receiving a stable dose for at least 6 months prior to screening
* If hydroxyurea treatment has been discontinued, at least 3 months have elapsed since last dose
* If transfusion in the 4 months prior to screening, then HbA level < 20% at screening
* Average of the initial two HbF levels ≥ 2.0 % within ≤ 7 days prior to the initial dose of HQK-1001. The two must be obtained ≥ 24 hours apart
* Ability to swallow tablets
* Able and willing to give informed consent and assent (if applicable)
* If subject is a woman of child-bearing potential (WCBP), she must have a negative serum pregnancy test within 7 days of first dose of HQK-1001
* If a subject is a WCBP, she must agree to use an effective form of contraception within 7 days of the initial dose of HQK-1001 and for one month after HQK-1001 discontinuation
* Sexually active male subjects (with WCBP partners) must agree to use latex condoms or ensure that their partner(s) use an effective form of contraception
* In the view of the Investigator, subject is able and willing to comply with necessary study procedures

Exclusion Criteria:

* More than 4 hospitalizations for acute sickle cell related events in the previous 12 months prior to screening
* Pulmonary hypertension requiring oxygen therapy
* QTc > 450 msec (male) or 470 msec (female) on screening ECG (QT corrected by Fridericia's formula)
* Assigned to a regular transfusion program
* Use of erythropoiesis stimulating agents within 90 days of screening
* ALT > 3x upper limit of normal (ULN)
* Serum creatinine > 1.2 mg/dL
* A serious, concurrent illness that would limit ability to complete or comply with the study requirements
* An acute vaso-occlusive event within 3 weeks prior to screening
* Creatine phosphokinase (CK) > 20% above the ULN
* An acute illness (e.g., febrile, GI, respiratory) within 72 hours prior to screening
* History of syncope, clinically significant dysrhythmias or resuscitation from sudden death
* Chronic opiate use, which, in the view of the Investigator, could confound evaluation of an investigational drug
* Current abuse of alcohol or drugs
* Received another investigational agent within 4 weeks or 5 half-lives, whichever is longer, prior to screening
* Currently pregnant or breast feeding a child
* Known infection with HIV-1
* Infection with hepatitis B or hepatitis C, such that patients are currently on therapy or will be placed on therapy during the trial

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety | Day 1 through Week 30
  Physical exams, vital signs, clinical laboratory safety assessments, ECG and adverse event monitoring.

SECONDARY OUTCOMES:
Fetal hemoglobin levels | Day 1 and Weeks 4, 8, 12, 16, 20, 25, 26 and 30
Incidence of sickle cell crisis events | Day 1 through Week 30

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ghalie, MD, MBA, Study Director — HemaQuest Pharmaceuticals Inc.
Locations (16):
- United States (9):
  - Children's Hospital and Research Center - Oakland, Oakland, California
  - University of Miami Miller School of Medicine - Dept of Pediatrics, Miami, Florida
  - Georgia Health Sciences University - Adult SIckle Cell Center, Augusta, Georgia
  - University of Illinois at Chicago - Dept of Pediatrics, Chicago, Illinois
  - LSU Health Sciences Center - Feist Weiller Cancer Center, Shreveport, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - University of North Carolina at Chapel Hill - Comprehensive Sickle Cell Program, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Univerisity of Texas Southwestern Medical Center at Dallas - Pediatric Hematology Oncology, Dallas, Texas
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - University Health Network Toronto General Hospital, Toronto, Ontario
- Abu El Reesh Pediatric University Hospital, Cairo, Egypt
- University of the West Indies - Sickle Cell Unit, Mona, Kingston, Jamaica
- Lebanon (3):
  - American University of Beirut Medical Center, Beirut
  - Rafik Hariri University Hospital, Beirut
  - Chronic Care Center, Hazmiyeh

REFERENCES:
- [Derived] Kutlar A, Reid ME, Inati A, Taher AT, Abboud MR, El-Beshlawy A, Buchanan GR, Smith H, Ataga KI, Perrine SP, Ghalie RG. A dose-escalation phase IIa study of 2,2-dimethylbutyrate (HQK-1001), an oral fetal globin inducer, in sickle cell disease. Am J Hematol. 2013 Nov;88(11):E255-60. doi: 10.1002/ajh.23533. Epub 2013 Oct 3. PMID 23828223